CLINICAL TRIAL: NCT05803187
Title: A Prospective, Observaional Multi-Center Phase IV Study to Evaluate the Efficacy and Safety of QLETLI (Adalimumab Biosimilar) in Pediatric and Juvenile Subjects With Severe Plaque Psoriasis (PISCES Trials)
Brief Title: Clinical Study of Stage IV Psoriasis in Children With Geleli
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: BAT-1406-008-CR
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter, prospective, observational phase IV clinical study. A total of 80 children and adolescents with severe plaque psoriasis were included in the study. The study is expected to last for 24 weeks (169 days). This study will evaluate the efficacy and safety of Valerie ® (Adalimumab Injection) in Chinese children over 4 years old and adolescents with severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. ) Patients and / or patient guardians voluntarily participated in the study and signed informed consent
2. )Age ≥ 4 years and < 18 years, male or female
3. ) The weight of patients should be 15 kg or more
4. ) Patients diagnosed with plaque psoriasis for at least 6 months ; at the same time, the researchers clarified the diagnosis of psoriasis
5. ) Patients with poor efficacy or unsuitable for local treatment and / or phototherapy
6. ) For patients with severe plaque psoriasis, the definition should meet one of the following conditions : Psoriasis static clinician overall assessment PGA score ≥ 4 points The body surface area of psoriatic lesions was BSA > 10 %. Psoriasis area and severity index PASI > 12 Children 's skin disease quality of life index ( CDLQI ) score > 10 points.

Exclusion Criteria:

1. A history of severe allergies or allergic reactions to monoclonal antibodies
2. Active infectious diseases ( including tuberculosis, hepatitis B, AIDS, syphilis, etc. )
3. Conform to any of the following criteria associated with latent or active TB infection :

   A history of active TB ≤3 years prior to screening (but if > 3 years, and a history of complete treatment Piece record, can also be grouped) During the screening period, there were signs or symptoms indicating active TB during medical history and / or physical examination ; recent close contact with people with active tuberculosis ( TB ) ; At the time of screening the interferon gamma release test tested positive if the subject's first interferon If the gamma release test results are inconclusive, the subject is excluded from the study;For subjects who have completed appropriate standard treatment for latent TB prior to screening and have no additional risk factors, radiographic findings or support for specific signs of latent or active TB,Possible for positive or inconclusive results. Exceptions will be made. The investigator will need to consult with a qualified infectomist to determine the risk of TB (including extra-pulmonary) and Discuss and decide with the sponsor;
4. Two pairs of hepatitis B surface antigen ( HBsAg ) were positive in screening. Or HBsAg negative, HBcAb positive and HBV-DNA positive.
5. There are serious, progressive or uncontrollable kidney, liver, blood, gastrointestinal, lung, heart blood. Tube, nerve or brain disease symptoms.
6. Patients received anti-tumor necrosis factor ( TNF ) or other biological agents with potential therapeutic effects on psoriasis within the previous 12 weeks.
7. Patients received intravenous anti-infective therapy within 30 days or oral anti-infective therapy within 14 days.
8. Local glucocorticoids, vitamin D derivatives, retinoic acid, calcineurin inhibitors ( TCI ) and other topical preparations with pharmacologically active ingredients were received within 7 days.
9. Local or UVB phototherapy within 7 days or psoralen or psoralen combined with ultraviolet A ( UVA ) phototherapy within 14 days.
10. Systemic treatment with non-biological agents for psoriasis including methotrexate, retinoic acids, cyclosporine, apulmiast, azathioprine, hydroxyurea, leflunomide, mexicophenol ester, sulfadiazine, calcineurase inhibitors, 6⁃ thiguanine for 14 days prior to baseline
11. Those who received any live vaccine within 3 months prior to receiving the first dose of the study drug, or during the study period.
12. Patients with erythrodermic psoriasis, pustular psoriasis, drug-induced or aggravated psoriasis, and newly minted guttate psoriasis
13. Patients who were judged unsuitable for inclusion by other investigators

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 80 children and adolescents with severe plaque psoriasis were enrolled in this study. Selected recipient Candidates must meet all inclusion criteria and not meet any exclusion criteria. Before performing any specific evaluation or Prior to the procedure, all subjects and/or guardians must sign written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Psoriasis lesion area and severity index (PASI) | Week 16 after administration
  Proportion of patients with a 75% decrease in PASI score at week 16 compared to baseline
Physician Global Assessment (PGA) | Week 16 after administration
  Proportion of patients with a PGA score of 0 ( clearance ) or 1 ( very mild ) at week 16

CONTACTS AND LOCATIONS:
Overall Officials: Jun Gu, Senior, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China